CLINICAL TRIAL: NCT06187727
Title: Clinical Study on Reducing Myocardial Infarction Siez After Primary PCI in Patients With ST Segment Elevation Myocardial Infarction by Using Henagliflozin
Brief Title: Henagliflozin Reducing Infarct Size After Priamry PCI in Patients With ST Segment Elevation Myocardial Infarction
Acronym: Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qian geng (Other)
Responsible Party: Sponsor-Investigator, Qian geng, MD, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Henagliflozin for infarction; Z-2017-26-2202-04 (Other Grant/Funding Number: China International Medical Fundinging)
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction; Heart Failure
Keywords: myocardial infartction; Ventricular remodeling
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Ventricular Remodeling | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- henagliflozein group (Experimental): Patients in henagliflozein group was given henagliflozein once a day for 6 months after myocardial infarction.
  Interventions: Drug: Henagliflozin
- Placebo group (No Intervention): Patients in placebo group was given palcebo once a day for 6 months after myocardial infarction.

INTERVENTIONS:
Drug: Henagliflozin — After primary PCI, Henggliflozin or Placebo was administered within 24 hours, followed by daily oral administration until 6 months post-acute myocardial infarction.
  Arms: henagliflozein group

SUMMARY:
This Randomized controlled intervention study recruited patients diagnosed with ST-segment elevation myocardial infarction (STEMI). A total of 240 patients were enrolled in either Henagliflozin group or control group. Patients in Henggliflozin group will be given by oral administration of Henggliflozin for 6 months post acute myocardial infarction. Prior to procedure, dynamic changes in myocardial enzymes were monitored. Major cardiovascular events, including non-fatal myocardial infarction, all-cause death, revascularization due to angina, and hospitalization for acute heart failure. This study aims to assess the impact of Henggelizin intervention on the reduction of myocardial infarction size (evaluated by cardiac enzyme) and improvement of left ventricular remodeling in patients with ST-segment elevation myocardial infarction.

DETAILED DESCRIPTION:
This Randomized controlled intervention study recruited patients diagnosed with ST-segment elevation myocardial infarction (STEMI) who were scheduled to undergo emergency percutaneous coronary intervention (PCI) . A total of 240 patients were selected for both the Henagliflozin group and control group. In the emergency room, clinical data would be collected, along with peripheral venous blood samples for laboratory examination. This examination should include blood routine analysis, myocardial enzyme, blood glucose levels, liver and kidney function, and brain natriuretic peptide precursor (NT proBNP) measurement. After primary PCI, Henggliflozin was administered, followed by daily oral administration of one tablet until 6 months post-acute myocardial infarction. Prior to procedure, dynamic changes in myocardial enzymes and electrocardiogram were monitored, with subsequent monitoring at 6 hours, 24 hours, and 48 hours after myocardial infarction. Perioperative complications were documented, followed by cardiac ultrasound assessments of myocardial wall motion and cardiac structure at seven days post primary PCI and six months post procedure. Major cardiovascular events, including non-fatal myocardial infarction, all-cause death, revascularization due to angina, and hospitalization for acute heart failure, were observed through follow-up at 1 month, 2 months, 3 months, and 6 months after PCI. This study aims to assess the impact of postoperative Henggelizin intervention on the reduction of myocardial infarction size and improvement of left ventricular remodeling in patients with ST-segment elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

1. STEMI patients with clear diagnosis: ischemic chest pain lasting for more than 30 minutes and adjacent to two or more leads of ST Segment elevation (limb lead ≥ 0.1mV, chest lead ≥ 0.2mV) with or without elevated myocardial enzyme levels;
2. Chest pain lasting less than 12 hours;
3. Age range from 18 to 80 years old;
4. Plans to undergo primary PCI ;
5. Informed consent form

Exclusion Criteria:

1. Mechanical complications;
2. Cardiogenic shock;
3. Experienced myocardial infarction within 6 months;
4. Aortic dissection;
5. Suffering from malignant tumors, severe liver and kidney failure, respiratory failure, or other short-term progressive diseases that researchers believe cannot be included
6. Urinary system infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of myocardial enzymes (CK-MB) | 3 days after the primary PCI
  Postoperative dynamic monitoring of myocardial enzyme （CK-MB）changes post infarction

SECONDARY OUTCOMES:
Left ventricular remodeling | 6 months after primary PCI
  Left ventricular remodeling evaluated by echocardiography，left ventricular end diastolic volume increase more than 20% compared bybaseline
contrast induced by nephropathy | 5 days after the primary PCI
  absolute increase in serum creatinine (SCr) 48-72 hours after primary PCI > 0.5 mg/dl or a relative increase > 25% compared with baseline SCr.
Cardiovascular adverse events | 12 months after primary PCI
  readmission due to heart failure, daeath, myocardial infarction
renal function renal function Renal function | 6 months after primary PCI
  Glomerular filtration rate evaluated glomerular filtration rate 6 months after primary PCI
Infarct size | 7 days after the primary PCI
  Infarct size measured by cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bai, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee TM, Chang NC, Lin SZ. Dapagliflozin, a selective SGLT2 Inhibitor, attenuated cardiac fibrosis by regulating the macrophage polarization via STAT3 signaling in infarcted rat hearts. Free Radic Biol Med. 2017 Mar;104:298-310. doi: 10.1016/j.freeradbiomed.2017.01.035. Epub 2017 Jan 26. PMID 28132924
- [Result] Tanajak P, Sa-Nguanmoo P, Sivasinprasasn S, Thummasorn S, Siri-Angkul N, Chattipakorn SC, Chattipakorn N. Cardioprotection of dapagliflozin and vildagliptin in rats with cardiac ischemia-reperfusion injury. J Endocrinol. 2018 Feb;236(2):69-84. doi: 10.1530/JOE-17-0457. Epub 2017 Nov 15. PMID 29142025
- [Result] Mizuno M, Kuno A, Yano T, Miki T, Oshima H, Sato T, Nakata K, Kimura Y, Tanno M, Miura T. Empagliflozin normalizes the size and number of mitochondria and prevents reduction in mitochondrial size after myocardial infarction in diabetic hearts. Physiol Rep. 2018 Jun;6(12):e13741. doi: 10.14814/phy2.13741. PMID 29932506
- [Result] Andreadou I, Efentakis P, Balafas E, Togliatto G, Davos CH, Varela A, Dimitriou CA, Nikolaou PE, Maratou E, Lambadiari V, Ikonomidis I, Kostomitsopoulos N, Brizzi MF, Dimitriadis G, Iliodromitis EK. Empagliflozin Limits Myocardial Infarction in Vivo and Cell Death in Vitro: Role of STAT3, Mitochondria, and Redox Aspects. Front Physiol. 2017 Dec 19;8:1077. doi: 10.3389/fphys.2017.01077. eCollection 2017. PMID 29311992
- [Result] Stone GW, Selker HP, Thiele H, Patel MR, Udelson JE, Ohman EM, Maehara A, Eitel I, Granger CB, Jenkins PL, Nichols M, Ben-Yehuda O. Relationship Between Infarct Size and Outcomes Following Primary PCI: Patient-Level Analysis From 10 Randomized Trials. J Am Coll Cardiol. 2016 Apr 12;67(14):1674-83. doi: 10.1016/j.jacc.2016.01.069. PMID 27056772